CLINICAL TRIAL: NCT06473272
Title: A Multi-center Prospective Cohort Study on the Evaluation of Vulnerability of Carotid Artery Plaques and Prediction of Cardio-Cerebrovascular Event Risk Using Ultrasonic Imaging
Brief Title: Evaluation of Vulnerability of Carotid Plaques and Prediction of Cardio-Cerebrovascular Event Using Ultrasonic Imaging
Status: Recruiting | Type: Observational
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Rong Wu, Principal Investigator, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: Shanghai1st-WR
Record Dates: First submitted 2024-06-04; First posted 2024-06-25 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Carotid Plaque; Ischemic Stroke; Cardiovascular Events
MeSH Terms: conditions — Ischemic Stroke | interventions — Blood Circulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Symptomatic group: The symptomatic group consisted of patients who were diagnosed with their first ipsilateral ischemic lesions in the carotid territory (anterior circulation) based on head computed tomography (CT) or magnetic resonance imaging (MRI) conducted within the previous 8 weeks.
  Interventions: Other: Cardiovascular and cerebrovascular diseases
- Asymptomatic group: The asymptomatic group included patients who showed no intracranial ischemic lesions on head CT/MRI images and exhibited no neurological symptoms.

INTERVENTIONS:
Other: Cardiovascular and cerebrovascular diseases — Cardiovascular and cerebrovascular diseases
  Groups: Symptomatic group

SUMMARY:
This study included patients with carotid artery atherosclerotic plaques to conduct multimodal ultrasound examinations, aiming to establish a plaque vulnerability assessment model based on ultrasonic imaging indicators, clinical history, and laboratory indicators. Based on the occurrence of cardiovascular and cerebrovascular events during the 3-year follow-up period, the correlation between the vulnerability of carotid plaques and the occurrence of cardiovascular and cerebrovascular events was explored. Furthermore, a cardiovascular and cerebrovascular risk prediction model for patients with plaques was established by combining multi-dimensional data indicators such as patients' clinical data and ultrasonic multimodal imaging data, forming a risk warning tool suitable for clinical use and providing a reference for risk management in patients with carotid artery plaques.

Research Objectives：

1. To establish a plaque vulnerability assessment model based on ultrasonic imaging indicators of plaques, clinical indicators of patients, and laboratory indicators.
2. To establish a cardiovascular and cerebrovascular risk prediction model for patients with carotid plaques by combining clinical indicators of patients and ultrasonic multimodal imaging data.
3. To screen ultrasonic imaging indicators for predicting cardiovascular and cerebrovascular events.

DETAILED DESCRIPTION:
This study is a prospective multi-center cohort study that aims to collect 600 patients with carotid artery plaques (including over 66,000 multimodal ultrasound image data), with patients coming from five participating centers. Starting from the collection of cases, the follow-up period is 36 months, during which the occurrence of cardiovascular and cerebrovascular events in patients will be observed. The relationship between multimodal ultrasonic imaging indicators, the vulnerability of carotid plaques, and cardiovascular and cerebrovascular events will be explored. Based on this, a cardiovascular and cerebrovascular risk prediction model for patients with carotid artery plaques will be established, forming a risk warning tool suitable for clinical use.

Inclusion criteria:

1. Patients who fully understand the purpose and significance of this experiment, voluntarily participate, and voluntarily sign the informed consent form;
2. Patients over 40 years old;
3. Patients with carotid plaque thickness ≥ 1.5 mm on conventional ultrasound, undergoing routine duplex ultrasound, contrast-enhanced ultrasound, ultrasound elastography, and three-dimensional ultrasound imaging.

Exclusion criteria:

1. Patients with severe cardiopulmonary insufficiency; allergy to sulfur hexafluoride; pregnant or lactating women; those with advanced tumors;
2. Poor quality of ultrasound images;
3. Patients who have previously undergone carotid artery stenting or endarterectomy on the same side as the carotid plaque.

The study aims to complete the establishment of an imaging database for 600 patients undergoing ultrasound examinations for carotid artery plaques, follow them up for 36 months, and record whether cardiovascular and cerebrovascular diseases occur.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who fully understand the purpose and significance of this experiment, voluntarily participate, and voluntarily sign the informed consent form;
2. Patients over 40 years old;
3. Patients with carotid plaque thickness ≥ 1.5 mm on conventional ultrasound, undergoing routine duplex ultrasound, contrast-enhanced ultrasound, ultrasound elastography, and three-dimensional ultrasound imaging.

Exclusion Criteria:

1. Patients with severe cardiopulmonary insufficiency; allergy to sulfur hexafluoride; pregnant or lactating women; those with advanced tumors;
2. Poor quality of ultrasound images;
3. Patients who have previously undergone carotid artery stenting or endarterectomy on the same side as the carotid plaque.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with carotid plaque
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
IPN semi-quantitative grading | 36 months
  Grade 0: no microbubbles seen within the plaque; Grade 1: microbubbles limited to the plaque shoulder or adventitial surface; Grade 2: microbubbles visible at the thickest part of the plaque, the intimal surface, or extensive enhancement within the plaque

SECONDARY OUTCOMES:
Plaque volume (mm^3) | 36 months
  using the software package provided with the ultrasound machine or post-processing software
Average shear wave velocity | 36 months
  After obtaining a stable grayscale image, select the shear wave elastography (SWE) mode and adjust the region of interest (ROI) to include the entire plaque. During the examination, ensure that the probe only has minimal contact with the skin to minimize compression artifacts. Freeze the image after stabilization, acquire the elastography image, and use the tracking tool to accurately outline the plaque boundary to obtain the average shear wave velocity (SWV).
Ulceration and low-echo regions (if present) | 36 months
  The largest area of surface ulceration and low-echo regions within the plaque

CONTACTS AND LOCATIONS:
Overall Officials: Rong Wu, Dr, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-30): https://cdn.clinicaltrials.gov/large-docs/72/NCT06473272/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-30): https://cdn.clinicaltrials.gov/large-docs/72/NCT06473272/ICF_001.pdf